CLINICAL TRIAL: NCT01966575
Title: Effect of Progestin-Induced Endometrial Shedding on Ovulation Induction Cycles With Clomiphene Citrate: A Randomized Study
Brief Title: Effect of Progestin-Induced Withdrawal Bleed on Ovulation Induction Cycles With Clomiphene Citrate
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Recent findings suggest that letrozole may be a superior Clomiphene Citrate.
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H13-02187
Record Dates: First submitted 2013-09-17; First posted 2013-10-21 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Polycystic Ovary Syndrome; Infertility
Keywords: Polycystic ovary syndrome; Progestin; Endometrial shedding; Ovulation induction cycles; Clomiphene citrate; Clinical pregnancy rate
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Progestins; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No withdrawal bleed (Experimental): No progestin prior to ovulation induction with clomiphene citrate
  Interventions: Drug: Progestin
- Withdrawal Bleed (No Intervention): Progestin prior to beginning ovulation induction with clomiphene citrate (standard care)

INTERVENTIONS:
Drug: Progestin — The experimental group will have no progestin prior to ovulation induction with clomiphene citrate, while the comparison group will have progestin medication prior to ovulation induction with clomiphene citrate, as per usual care.
  Other Names: medroxyprogesterone acetate (MPA), i.e. Provera
  Arms: No withdrawal bleed

SUMMARY:
Women with polycystic ovary syndrome (PCOS) can suffer from infertility because they do not produce an egg each month, resulting in irregular periods. As a result, these women often need a medication called clomiphene citrate (clomiphene) to induce ovulation. A traditional 'clomiphene protocol' begins with a short course of progestin treatment to bring on a period (termed a 'withdrawal bleed') before starting the clomiphene medication. Newer evidence, however, has suggested that this progestin-induced shedding of the uterine lining (i.e., withdrawal bleed) may decrease the chances of pregnancy. The purpose of our study is to determine whether withdrawal bleeding has an impact on pregnancy rates for patients with PCOS undergoing a clomiphene cycle.

It is hypothesized that patients who undergo ovulation induction with clomiphene citrate without prior endometrial shedding will have higher clinical pregnancy rates than those who begin with a progestin-induced withdrawal bleed.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome (Rotterdam 2003 Consensus Criteria) and a diagnosis of anovulatory infertility
* Age 18-38 years
* At least 1 patent fallopian tube (as demonstrated by hysterosalpingogram, hydrotubation or hysterosonogram within the last year)
* Normal semen analysis (total motile sperm count >20million/ml)
* Normal uterine cavity (as demonstrated by hysterosalpingogram, hydrotubation or hysterosonogram within the last year)
* Undergoing ovulation-induction with clomiphene citrate without intra-uterine insemination (IUI)

Exclusion Criteria:

* Body mass index (BMI) < 17 kg/m2 or > 40 kg/m2
* Prior treatment with clomiphene citrate
* Presence of a hydrosalpinx (as seen on ultrasound, hysterosalpingogram, hydrotubation or hysterosonogram)
* Those with systemic disease such as diabetes mellitus, uncontrolled thyroid disease, systemic lupus erythematosus and antiphospholipid antibody syndrome
* Any other cause of infertility other than anovulation

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate per ovulation | 6 weeks after starting clomiphene
  clinical pregnancy rate (gestational sac seen on ultrasound approximately 6-7 weeks after starting clomiphene) per ovulation

SECONDARY OUTCOMES:
cumulative pregnancy rate | assessed 9 months after the ovulation induction cycles
  cumulative pregnancy rate
ovulation rate | assessed 1 month after each induced ovulation cycle
  ovulation rate (progesterone >10nmol/L per clomiphene cycle)
ongoing pregnancy rate | assessed 12 weeks after clinical pregnancy is acheived
  ongoing pregnancy rate (pregnancy with a fetal heartbeat >12 weeks gestational age)
miscarriage rate | Assessed 4 months after clinical pregnancy acheived
  miscarriage rate
multiple pregnancy rate | Assessed 4 months after clinical pregnancy acheived
  multiple pregnancy rate (twins and higher order multiples)
endometrial thickness | Assessed at 1 month after conception
  endometrial thickness (assessed via transvaginal ultrasound)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Havelock, MD, Principal Investigator — University of British Columbia
Locations (1):
- Pacific Centre for Reproductive Medicine, Burnaby, British Columbia, Canada